CLINICAL TRIAL: NCT04065087
Title: A Phase 1/2, Randomized, Placebo-controlled Study to Evaluate Safety, Tolerability, Anti-tumor Activity of GX-I7 Plus Adjuvant Temozolomide Combination Regimen in Patients With Newly Diagnosed With Glioblastoma
Brief Title: Efficacy and Safety Study of GX-I7 Plus Adjuvant Temozolomide Combination in Patients With Newly Diagnosed Glioblastoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Canceled by the sponsor
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GX-I7-CA-007
Record Dates: First submitted 2019-07-25; First posted 2019-08-22 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Newly Diagnosed Glioblastoma
MeSH Terms: interventions — efineptakin alfa

STUDY DESIGN:
Intervention Model Description: Phase 1: sequential dose escalation Phase 2: randomized, placebo controlled, parallel arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GX-I7 (Experimental): GX-I7 administered until Progression of Disease
  Interventions: Biological: GX-I7
- Placebo (Placebo Comparator): Placebo administered until Progression of Disease
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: GX-I7 — Investigational drug
  Arms: GX-I7
Other: Placebo — Placebo drug
  Arms: Placebo

SUMMARY:
This is a phase 1/2, randomized, placebo-controlled study to evaluate safety, tolerability, anti-tumor activity and impact on absolute lymphocyte count of GX-I7 plus adjuvant temozolomide combination regimen in patients with newly diagnosed with glioblastoma who completed standard concurrent chemo-radiation therapy (CCRT)

DETAILED DESCRIPTION:
In dose escalation stage (Phase 1 part), low/intermediate/high dose of GX-I7 will be administered in combination with adjuvant temozolomide to find recommended phase 2 dose.

Phase 2 part will be randomized, placebo controlled study and GX-I7 or Placebo will be administered in combination with adjuvant temozolomide treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF)
2. Age ≥ 19 years
3. Gross total resection equal to or greater than 80% based on post-op MRI, compared to pre-op MRI (Patients requiring biopsy only is not eligible)
4. Patients newly diagnosed with glioblastoma either by imaging or pathology testing, requiring concurrent chemo-radiotherapy (CCRT) and adjuvant temozolomide chemotherapy with curative intent
5. Karnofsky score ≥ 60
6. Life expectancy > 12 weeks

Exclusion Criteria:

1. Gliomatosis cerebri
2. Isocitrate dehydrogenase 1 & 2 mutation
3. Pregnant or breast feeding women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-22 (Estimated); Primary Completion 2022-05-27 (Estimated); Study Completion 2022-08-27 (Estimated)

PRIMARY OUTCOMES:
lymphocyte count | 12 weeks
  Change in absolute lymphocyte count

SECONDARY OUTCOMES:
Overall survival | 36 months
  Median overall survival
Progression free survival | 24 months
  Median progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent Hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No